CLINICAL TRIAL: NCT02407171
Title: A Phase I/II Trial of Evaluating the Combination of MK-3475 and Stereotactic Body Radiotherapy in Patients With Metastatic Melanoma or NSCLC
Brief Title: Evaluating the Combination of MK-3475 and Sterotactic Body Radiotherapy in Patients With Metastatic Melanoma or NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1411014879
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Melanoma; Lung Cancer
MeSH Terms: conditions — Melanoma; Lung Neoplasms | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Non Small Cell Lung Cancer, Phase I (Experimental): Dose escalation cohort for patients with Non Small Cell Lung Cancer (NSCLC). The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.
  Interventions: Drug: MK-3475; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Non-Lung, Phase I (Experimental): Dose escalation cohort for non lung cancer patients. The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.
  Interventions: Drug: MK-3475; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Melanoma Expansion Cohort (Experimental): Phase 2a expansion cohort for patients with melanoma. Patients will be treated at the maximum tolerated dose discovered in phase I.
  Interventions: Drug: MK-3475; Radiation: Stereotactic Body Radiation Therapy (SBRT)
- Non Small Cell Lung Cancer Expansion Cohort (Experimental): Phase 2a expansion cohort for patients with NSCLC. Patients will be treated at the maximum tolerated dose discovered in phase I.
  Interventions: Drug: MK-3475; Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: MK-3475 — 200 mg every 2 weeks by IV infusion
Radiation: Stereotactic Body Radiation Therapy (SBRT) — The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).

SUMMARY:
This is a 2-part prospective trial examining the ability of Stereotactic Body Radiation Therapy (SBRT) to induce a response to MK-3475, a humanized antibody to PD-1, in patients who progress on this antibody. Patients with metastatic melanoma will be enrolled after they have progressed on anti-PD-1 therapy. Patients with metastatic NSCLC (previously untreated with anti-PD-1 or anti-PD-L1 therapy) will be enrolled and treated with MK-3475 until they exhibit progression of disease. At this point (when patients have demonstrated progression of disease) a single target lesion will be selected and treated with SBRT, and then MK-3475 will be restarted and continued until there is further progression of disease. The first phase of the study is a radiation dose escalation with a constant dose of MK-3475. The second part of the study includes expansion cohorts of NSCLC and melanoma patients.

DETAILED DESCRIPTION:
The phase 1b portion of the trial is a radiation dose escalation study to determine the maximum tolerated dose (MTD) of SBRT when given to patients previously and subsequently exposed to MK-3475. Because the class of PD-1 inhibitory antibodies conveys a risk of pneumonitis, there will be two parallel dose escalation arms- Arm A will include SBRT targets in the lung parenchyma, and Arm B will be limited to targets outside the lung parenchyma. Each arm will be separately escalated, and two MTDs will be determined. The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.

The phase 2a portion of the study includes 2 expansion cohorts, for melanoma and NSCLC, with SBRT delivered at the MTD. The primary endpoint of this phase of the study is the overall response rate to post-SBRT MK-3475. Secondary endpoints include determining the time to progression, overall survival, and exploratory biomarkers.

IND exempt per FDA.

Inclusion/Exclusion Criteria Updated 4/7/2016

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Have metastatic melanoma or NSCLC, or locally advanced NSCLC not suitable for curative-intent local therapy.
* For melanoma patients and NSCLC patients treated with prior anti-PD-1 therapy, patients must have received prior PD-1 therapy and have progressed (irPD) by irRC.
* Have 2 or more measurable sites of disease as defined by either RECIST 1.1, or cutaneous lesions at least 1 cm in greatest dimension
* Have at least one site of disease that is considered potentially suitable for treatment with SBRT
* Have provided tissue from an archival or newly obtained tissue sample of a tumor lesion, sufficient for analysis of PD-L1 and other biomarkers. Patients who have had PD-L1 analysis previously performed at Merck can substitute earlier analysis results and are not required to submit additional tissue for PD-L1 testing. Expression of PD-L1 is NOT required for study entry.
* Have a performance status of 0, 1 or 2 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 28 days of protocol treatment.

Table 1. Adequate Organ Function Laboratory Values (System/Laboratory Value)

Hematological

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥100,000 / mcL
* Hemoglobin ≥9 g/dL

Renal

* Measured or calculated creatinine** clearance ≤1.5 X upper limit of normal (ULN)
* (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic
* Serum total bilirubin ≤ 1.5 X ULN OR
* Direct bilirubin Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases

  **(Creatinine clearance should be calculated per institutional standard. )
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Has had radiation therapy within 2 weeks of the first protocol treatment.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 2 weeks of the first protocol treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 weeks of the first protocol treatment. The use of low-dose steroids for management of chronic conditions is allowed.
* Non-small cell lung cancer patients enrolling to MK-3475 as first protocol therapy (no prior anti-PD-1 therapy): Has had a prior monoclonal antibody within 4 weeks prior to first protocol treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks of the first protocol treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: Patients who have had prior treatments with Tyrosine Kinase Inhibitors (e.g. Tarceva) require only a 72-hour washout period prior to starting protocol treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active and untreated brain (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an example of an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Those with a history of hypothyroidism who are now stable on hormone replacement will not be excluded. Those with Sjorgen's syndrome will not be excluded from the study.
* Has a history of (non-infectious) pneumonitis that required steroids, current pneumonitis or evidence of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Campbell, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy: Participants with no prior PD-1 therapy that began in the Phase 1: Lung Targets + MK-3475 and then moved to Phase 2 NSCLC phase of the study.
- Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD: Participants previously treated with immunotherapy/irPD that began in the Phase 1: Lung Targets + MK-3475 and then moved to Phase 2 NSCLC phase of the study.
- Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy: Participants no prior PD-1 therapy that began in the Phase 1: Non-Lung Target + MK-3475 and then moved to Phase 2 melanoma phase of the study.
- Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD: Participants previously treated with immunotherapy/irPD that began in the Phase 1: Non-Lung Target and then moved to Phase 2: melanoma phase of the study.
- Phase 2: NSCLC, no Prior PD-1 Therapy: Patients in this portion of Phase 2, NSCLC, no prior PD-1 therapy.
  Phase 2 ONLY patients
- Phase 2: NSCLC or Melanoma, Previously Treated With Immunotherpay, With irPD: Phase 2a expansion cohort for patients with melanoma. Patients will be treated at the maximum tolerated dose discovered in phase I.
  Drug: MK-3475 200 mg every 2 weeks by IV infusion
  Radiation: Stereotactic Body Radiation Therapy (SBRT) The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).
  Phase 2 ONLY patients
Period: Phase 1 Dose Escalation
Arm/Group | Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy | Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD | Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy | Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD | Phase 2: NSCLC, no Prior PD-1 Therapy | Phase 2: NSCLC or Melanoma, Previously Treated With Immunotherpay, With irPD
Started | 10 | 3 | 5 | 6 | 0 (Phase 2 ONLY patients) | 0 (Phase 2 ONLY patients)
Dose Escalation 30 GY3 | 3 | 3 | 4 | 3 | 0 | 0
Dose Escalation 30 GY5 | 7 | 0 | 1 | 3 | 0 | 0
Completed | 10 | 3 | 5 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Treatment
Arm/Group | Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy | Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD | Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy | Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD | Phase 2: NSCLC, no Prior PD-1 Therapy | Phase 2: NSCLC or Melanoma, Previously Treated With Immunotherpay, With irPD
Started | 10 | 3 | 5 | 6 | 35 | 2
Received SBRT | 10 | 3 | 5 | 6 | 0 | 2
Completed | 10 | 3 | 5 | 6 | 35 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for participants in the study arm in which they began the study. Phase 1 participants included in the Phase 2 portion are presented in a single arm as the enrollment numbers are presented combined overall for both Phases.
Groups:
- Phase 2: Pre-SBRT for NSCLC: Patients in this portion of Phase 2, never progressed to receive SBRT.
- Phase 2: EC: Melanoma With Prior PD1: Phase 2a expansion cohort for patients with melanoma. Patients will be treated at the maximum tolerated dose discovered in phase I.
  Drug: MK-3475 200 mg every 2 weeks by IV infusion
  Radiation: Stereotactic Body Radiation Therapy (SBRT) The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).
- Total: Total of all reporting groups
Arm/Group | Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy | Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD | Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy | Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD | Phase 2: Pre-SBRT for NSCLC | Phase 2: EC: Melanoma With Prior PD1 | Total
Number analyzed (Participants) | 10 | 3 | 5 | 6 | 35 | 2 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (13.7) | 74.3 (13.6) | 67.8 (6.7) | 59.5 (6.4) | 67.6 (10.5) | 65.0 (7.1) | 67.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 2 | 5 | 19 | 0 | 36
  Male | 2 | 1 | 3 | 1 | 16 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 3 | 5 | 6 | 32 | 2 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 10 | 3 | 4 | 6 | 32 | 2 | 57
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 3 | 5 | 6 | 35 | 2 | 60

OUTCOME MEASURES:

1. Primary Outcome: Phase 2, Overall Response
Description: Phase 2 primary endpoint is the overall response count of patients to post-SBRT MK-3475. Overall response was evaluated using Response Evaluation Criteria In Solid Tumors (RECIST). The following are counts of those that were assessed to have the following responses: Complete response (CR), Partial response (PR), Stable disease (SD), Progressive disease (PD), Not Evaluable.
Time Frame: up to 12 months
Population: Only those that received SBRT.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy: Dose escalation cohort for patients with Non Small Cell Lung Cancer (NSCLC). The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.
  MK-3475: 200 mg every 2 weeks by IV infusion
  Stereotactic Body Radiation Therapy (SBRT): The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).
- Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD; Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD: Dose escalation cohort for non lung cancer patients. The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.
  MK-3475: 200 mg every 2 weeks by IV infusion
- Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy: Dose escalation cohort for non lung cancer patients. The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.
  MK-3475: 200 mg every 2 weeks by IV infusion
  Stereotactic Body Radiation Therapy (SBRT): The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).
- Phase 2: NSCLC or Melanoma, no Prior PD-1 Therapy: Patients in this portion of Phase 2, NSCLC or melanoma, no prior PD-1 therapy.
  Phase 2 ONLY patients
- Phase 2: Melanoma, Previously Treated With Immunotherpay, With irPD: Phase 2a expansion cohort for patients with melanoma. Patients will be treated at the maximum tolerated dose discovered in phase I.
  Drug: MK-3475 200 mg every 2 weeks by IV infusion
  Radiation: Stereotactic Body Radiation Therapy (SBRT) The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).
  Phase 2 ONLY patients
Arm/Group | Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy | Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD | Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy | Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD | Phase 2: NSCLC or Melanoma, no Prior PD-1 Therapy | Phase 2: Melanoma, Previously Treated With Immunotherpay, With irPD
Number analyzed (Participants) | 10 | 3 | 5 | 6 | 0 | 2
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 1 | 0 | 0 | 0 | 0 | 0
  Stable disease (SD) | 4 | 0 | 2 | 2 | 0 | 1
  Progressive disease (PD) | 5 | 3 | 1 | 3 | 0 | 1
  Not Evaluable | 0 | 0 | 2 | 1 | 0 | 0

2. Primary Outcome: Phase 1, Dose-Limiting Toxicity
Description: Phase 1 primary endpoint will be the presence of a dose limiting toxicity. Maximum tolerated dose will be the highest dose at which there is not a dose limiting toxicity. This could be either 3000 cGy in 5 fractions or 3 fractions. Presented are counts of the maximum tolerated of participants per arm. Results are summarized by Lung or Non-Lung targets overall.
Time Frame: up to 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: SBRT Dose Esc. for Lung Targets + MK-3475: Dose escalation cohort for patients with Non Small Cell Lung Cancer (NSCLC). The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.
  MK-3475: 200 mg every 2 weeks by IV infusion
  Stereotactic Body Radiation Therapy (SBRT): The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).
- Phase 1: SBRT Dose Esc. Non-Lung Target + MK-3475: Dose escalation cohort for non lung cancer patients. The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction). If there is dose-limiting toxicity at the lowest cohort, that arm will be closed and SBRT to that site will be discontinued.
  MK-3475: 200 mg every 2 weeks by IV infusion
  Stereotactic Body Radiation Therapy (SBRT): The starting dose will be 3000 cGy in 5 fractions; there will be one dose escalation cohort (3000 cGy in 3 fractions), and if necessary one dose de-escalation cohort (1000 cGy in a single fraction).
Arm/Group | Phase 1: SBRT Dose Esc. for Lung Targets + MK-3475 | Phase 1: SBRT Dose Esc. Non-Lung Target + MK-3475
Number analyzed (Participants) | 13 | 11
Participants
  3000 cGy in 5 fractions | 7 | 4
  3000 cGy in 3 fractions | 6 | 7

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Adverse event reporting was collected at the patient level and is not split by phase 1/phase 2. The study completion was delayed for a number of reasons, including the health of the original principal investigator.
Groups:
- Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy: Dose escalation cohort for patients with Non Small Cell Lung Cancer (NSCLC). These participants then entered Phase 2 with no prior PD-1 therapy.
- Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD: Dose escalation cohort for Non Small Cell Lung Cancer (NSCLC) These participants then entered Phase 2 previously treated with immunotherapy/irPD.
- Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy: Dose escalation cohort for non lung cancer patients. These participants then entered Phase 2 with no prior PD-1 therapy.
- Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD: Dose escalation cohort for non lung cancer patients. These participants then entered Phase 2 previously treated with immunotherapy/irPD.
- Phase 2: NSCLC With no Prior PD-1 Therapy: Patients in this portion of Phase 2, NSCLC with no prior PD-1 therapy.
  Phase 2 ONLY patients
- Phase 2: Melanoma, Previously Treated With Immunotherpay, With irPD: Phase 2a expansion cohort for patients with melanoma- previously treated with immunotherapy/irPD.
  Phase 2(a) ONLY patients
Arm/Group | Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy | Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD | Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy | Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD | Phase 2: NSCLC With no Prior PD-1 Therapy | Phase 2: Melanoma, Previously Treated With Immunotherpay, With irPD
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/3 | 1/5 | 0/6 | 3/35 | 0/2
Serious Adverse Events (participants affected / at risk) | 5/10 | 0/3 | 1/5 | 1/6 | 13/35 | 0/2
Other Adverse Events (participants affected / at risk) | 10/10 | 3/3 | 5/5 | 6/6 | 35/35 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy (N=10) | Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD (N=3) | Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy (N=5) | Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD (N=6) | Phase 2: NSCLC With no Prior PD-1 Therapy (N=35) | Phase 2: Melanoma, Previously Treated With Immunotherpay, With irPD (N=2)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Lung Targets + MK-3475 / Phase 2 NSCLC, no Prior PD-1 Therapy (N=10) | Phase 1: Lung Targets / Phase 2: NSCLC, Previously Treated With Immunotherapy/irPD (N=3) | Phase 1: Non-Lung Target + MK-3475 / Phase 2 Melanoma, no Prior PD-1 Therapy (N=5) | Phase 1: Non-Lung Target / Phase 2: Melanoma, Previously Treated With Immunotherapy/irPD (N=6) | Phase 2: NSCLC With no Prior PD-1 Therapy (N=35) | Phase 2: Melanoma, Previously Treated With Immunotherpay, With irPD (N=2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight loss (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 1 (1) | 1 (2)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (2) | 1 (2) | 7 (10) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 8 (10) | 1 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 2 (3) | 4 (6) | 1 (1) | 20 (27) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 1 (2) | 2 (3) | 21 (23) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 10 (11) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (4) | 2 (2) | 4 (4) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 3 (3) | 8 (8) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (3) | 0 (0) | 1 (2) | 8 (14) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 8 (8) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye disorders - Other (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 4 (5) | 2 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 1 (1) | 2 (2) | 3 (3) | 11 (13) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (11) | 0 (0) | 1 (1) | 2 (3) | 9 (15) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (2) | 3 (6) | 6 (7) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (4) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (12) | 2 (2) | 5 (10) | 6 (6) | 26 (31) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (13) | 1 (1)
Pain (General disorders) | 7 (8) | 1 (1) | 3 (4) | 1 (1) | 13 (19) | 2 (4)
Edema limbs (General disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT02407171/Prot_SAP_000.pdf